CLINICAL TRIAL: NCT02832453
Title: Supervised Physical Exercise and Lifestyle Counselling in the Management of Metabolic Risk in Low-active Adults; a Controlled Randomized Trial. Belluga't de CAP a Peus
Brief Title: Metabolic Risk Management, Physical Exercise and Lifestyle Counselling in Low-active Adults; Controlled Randomized Trial
Acronym: BELLUGAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: INEFC-Lleida (Other)
Collaborators: Institut Català de la Salut (Other); Universitat de Lleida (Other); Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Principal Investigator, Assumpta Ensenyat, Dr Assumpta Ensenyat (MD, PhD) Exercise Physiology, INEFC-Lleida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-PINEFC00003
Record Dates: First submitted 2016-07-06; First posted 2016-07-14 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Metabolic Syndrome X; Lifestyle-related Condition; Lifestyle Risk Reduction; Cardiovascular Risk Factor
Keywords: High intensity physical exercise; Primary health care; Behaviour change interventions
MeSH Terms: conditions — Metabolic Syndrome; Mental Disorders; Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lifestyle counseling (Other): This group will receive lifestyle counselling but not supervised exercise training sessions
  Interventions: Behavioral: Lifestyle
- Aerobic interval training (Experimental): This group will receive lifestyle counselling plus supervised high intensity (80%VO2max) interval exercise training sessions
  Interventions: Behavioral: Lifestyle; Behavioral: Aerobic interval training
- Traditional continous training (Active Comparator): This group will receive lifestyle counselling plus supervised moderate intensity (60%VO2max) continous exercise training sessions
  Interventions: Behavioral: Lifestyle; Behavioral: Traditional continous training

INTERVENTIONS:
Behavioral: Lifestyle — The counselling program consists of 6 group meetings of 1 hour and 3 individual consultations of at least 15 minutes each. Sessions will be set up with the aim to enhance knowledge and empowerment related to physical activity, sedentary conducts, dietary habits, as well as strategies for behaviour change will be given. Individual consultations will focus on establishing realistic objectives and to involve the participants in taking decisions.
Behavioral: Aerobic interval training — The supervised aerobic interval training will consist of 16 supervised group training lessons lasting 60 minutes and 32 individual nonsupervised training lessons that would be self-administered by each participant. The main part of the training lessons will consist of 4 series of 4 minutes of cycling at a heart rate of 80% of the VO2peak interspersed with active pauses of 2 minutes at 60% of the VO2peak .
  Arms: Aerobic interval training
Behavioral: Traditional continous training — The supervised traditional continous training will consist of 16 supervised group training lessons lasting 60 minutes and 32 individual nonsupervised training lessons that would be self-administered by each participant. The main part of the training lessons will consist of activities such as walking, cycling, or tonification exercises always at an intensity of 60% of the VO2peak.
  Arms: Traditional continous training

SUMMARY:
The purpose of this study is evaluate the effectiveness of different doses of supervised exercise training intensity -concomitant to lifestyle counselling- as a Primary Health Care intervention tool for the management of the metabolic syndrome in low active adults with one or more metabolic risk factors.

Secondary aims of the study are to investigate the effects of these interventions on systemic inflammation and adipose tissue function, cardiorespiratory fitness, physical activity and sedentary habits, and the cost-effectiveness of the intervention with regard to health related quality of life.

The general hypothesis is that adults with risk factors for metabolic syndrome participating in interventions for the promotion of a healthy lifestyle that together with counselling strategies will include supervised physical exercise of vigorous intensity will present greater improvements in terms of metabolic risk, physical condition, physical activity/sedentary behaviours and psychological parameters at the end of the intervention and at 6-months follow-up than participants in interventions for the promotion of a healthy lifestyle that will include counselling plus physical exercise of low-to-moderate intensity or interventions based exclusively on counselling.

It is a three arms controlled randomized clinical trial implemented in the Primary Health Care setting and of 10 months duration.

DETAILED DESCRIPTION:
The purpose of this study is evaluate the effectiveness of different doses of supervised exercise training intensity -concomitant to lifestyle counselling- as a Primary Health Care intervention tool for the management of the metabolic syndrome in low active adults with one or more metabolic risk factors.

Secondary aims of the study are to investigate the effects of these interventions on systemic inflammation and adipose tissue function, cardiorespiratory fitness, physical activity and sedentary habits, and the cost-effectiveness of the intervention with regard to health related quality of life.

The general hypothesis is that adults with risk factors for metabolic syndrome participating in interventions for the promotion of a healthy lifestyle that together with counselling strategies will include supervised physical exercise of vigorous intensity will present greater improvements in terms of metabolic risk, physical condition, physical activity/sedentary behaviours and psychological parameters at the end of the intervention and at 6-months follow-up than participants in interventions for the promotion of a healthy lifestyle that will include counselling plus physical exercise of low-to-moderate intensity or interventions based exclusively on counselling.

It is a three arms controlled randomized clinical trial implemented in the Primary Health Care setting and of 10 months duration.

Adults aged 30 to 52 years with metabolic risk factors will be randomized in three intervention groups that will be given one of the following: assessment on healthy lifestyle plus high intensity physical exercise supervision (3 individual and 6 group sessions + 16 supervised training lessons); assessment plus low-to-moderate intensity physical exercise supervision (3 individual and 6 group sessions + 16 supervised training lessons) or assessment-based programme without physical exercise supervision (3 individual and 6 group sessions).

The main output variables evaluated will be: a) risk factors for the metabolic syndrome (waist circumference, blood pressure, and plasma triglycerides, high density lipoproteins and glucose), systemic inflammation and adipose tissue functionality, physical activity habits and sedentary conducts, dietary habits, quality of life related to health, self-efficacy and empowerment. The economic cost will also be analysed to determine the cost-effectiveness of the program. These variables will be assessed 3 times alongside the study: at baseline, at the end of the 4 months intervention, and at 6 months follow-up. It has been estimated to recruit 33 participants per group, which are 100 participants.

ELIGIBILITY:
Inclusion Criteria:

* Low active (achieving less than 150 minutes/week of moderate-to-vigorous physical activity or have not participated in any supervised exercise programs for at least the last 6 months).
* Having one or more risk factors for metabolic syndrome (Marcuello et al., 2013) (waist circumference >94.5 cm for men and >89.5 cm for women; blood pressure ≥130/85 mmHg; triglycerides in plasma ≥150 mg/dL; high density lipoprotein cholesterol in plasma <40 mg/dL for men and <50 mg/dL for women; fasting glycaemia ≥100 mg/dL).
* Accept and sign the written informed consent.
* Accept the randomized group assignment.

Exclusion Criteria:

* Couples or individuals living in the same house
* Morbid obesity (BMI ≥ 40).
* A past/current history and/or physical examination or laboratory findings of significant diseases of cardiovascular, respiratory, neuromuscular, psychiatric diseases/disorders.
* Diseases/disorders that may contraindicate performing physical exercise or a stress test.

Ages: 30 Years to 52 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2016-02; Primary Completion 2017-06 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in metabolic risc score | 3 time points: at baseline, 4 months (end of the intervention) and at 6 months after the end of the intervention.
  A continuous metabolic syndrome risk score (cMSSy) will be calculated as described by Wijndaele (Wijndaele et al., 2006). The score contains the five risk factors considered in the definition of the metabolic syndrome (Expert panel on detection, 2001; Marcuello et al., 2013), that is waist circumference, triglycerides, high density lipoproteins cholesterol, systolic blood pressure and plasma glucose.

SECONDARY OUTCOMES:
Change from baseline in cardiorespiratory fitness | 3 time points: at baseline, 4 months (end of the intervention) and at 6 months after the end of the intervention.
  Improvement of peak oxygen uptake (VO2peak). Cardiorespiratory fitness will be assessed by means of voluntary maximal graded exercise on a cycle ergometer while measuring oxygen consumption (VO2).
Change from baseline in active lifestyle | 3 time points: at baseline, 4 months (end of the intervention) and at 6 months after the end of the intervention.
  Daily time spent at moderate-to-vigorous physical activity. Participants will wear Actigraph accelerometers (GT3X+ models) during all day for seven consecutive days. Cut points for moderate-to-vigorous physical activity will be set above 2020 counts per minute.
Change from baseline in sedentary time | 3 time points: at baseline, 4 months (end of the intervention) and at 6 months after the end of the intervention.
  Reduction of the daily time devoted to sedentary conducts. Participants will wear Actigraph accelerometers (GT3X+ models) during all day for seven consecutive days. Cut points for sedentary conducts will be set under 100 counts per minute.
Change from baseline in dietary habits | 3 time points: at baseline, 4 months (end of the intervention) and at 6 months after the end of the intervention.
  Improvement of healthy eating index
Change from baseline in physical activity self-efficacy questionnaire | 3 time points: at baseline, 4 months (end of the intervention) and at 6 months after the end of the intervention.
  Spanish version of the physical activity scale (Fernández-Cabrera, Medina, Rueda, Ordoñez, & León, 2012)
Change from baseline in empowerment | 3 time points: at baseline, 4 months (end of the intervention) and at 6 months after the end of the intervention.
  Health Empowerment Scale (HES) (Serrani, 2014)
Change from baseline in health related quality of life at the end of the intervention | 3 time points: at baseline, 4 months (end of the intervention) and at 6 months after the end of the intervention.
  Quality of life questionaire (EQ-5D)
Change from baseline in health related quality of life | 3 time points: at baseline, 4 months (end of the intervention) and at 6 months after the end of the intervention.
  Quality of life questionaire (EQ-5D)
Change from baseline in interleucin-6 | 3 time points: at baseline, 4 months (end of the intervention) and at 6 months after the end of the intervention.
  Fasting blood samples will be drawn to determine interleukin by cytometry.
Change from baseline in adiponectin | 3 time points: at baseline, 4 months (end of the intervention) and at 6 months after the end of the intervention.
  Fasting blood samples will be drawn to determine adiponectin by cytometry.
Change from baseline in plasma metabolome | 3 time points: at baseline, 4 months (end of the intervention) and at 6 months after the end of the intervention.
  Fasting blood samples will be drawn to determine plasma metabolome.

OTHER OUTCOMES:
Cost-effectiveness of the intervention | 4 months
  Direct and indirect costs of setting and running the interventions will be collected for the economic evaluation analysis by means of questionnaires. HRQoL scores will be used to weight survival years and generate quality adjusted life years (QALYs ). The cost-effectiveness analysis will be conducted according to the current practice methods for economic evaluation (Frew et al., 2014).

CONTACTS AND LOCATIONS:
Overall Officials: Assumpta Ensenyat, MD, PhD, Principal Investigator — INEFC-Lleida
Locations (1):
- INEFC-Lleida, Lleida, Spain

IPD SHARING:
Plan to Share IPD: Undecided
At present we have not planned to share data. Probably at the end of the trail we will put them on the repository of the University of Lleida.

REFERENCES:
- [Derived] Ensenyat A, Espigares-Tribo G, Machado-Da-Silva L, Sinfreu-Bergues X, Blanco A. Semisupervised Physical Exercise and Lifestyle Counseling in Cardiometabolic Risk Management in Sedentary Adults: Controlled Randomized Trial (BELLUGAT). J Phys Act Health. 2020 Jun 12;17(7):744-755. doi: 10.1123/jpah.2019-0409. PMID 32531762
- [Derived] Ensenyat A, Espigares-Tribo G, Machado L, Verdejo FJ, Rodriguez-Arregui R, Serrano J, Miret M, Galindo G, Blanco A, Marsal JR, Sarriegui S, Sinfreu-Bergues X, Serra-Paya N. Metabolic risk management, physical exercise and lifestyle counselling in low-active adults: controlled randomized trial (BELLUGAT). BMC Public Health. 2017 Mar 14;17(1):257. doi: 10.1186/s12889-017-4144-8. PMID 28292282